CLINICAL TRIAL: NCT05087823
Title: Measurements of Lipoproteins, Apolipoproteins, and Lipids in Three Separate Oral Challenges - Fat, Sugar, and Mixed Test Meals
Brief Title: The Mixed Meal Challenge Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Thomas R. Ziegler, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00116934
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases; Hyperlipidemias
Keywords: Prevention; Hyperlipidemia; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipid, Glucose, and Mixed Meal Challenges (Experimental): Participants will take part in three different meal challenges on three separate days with approximately two weeks in between. The first meal challenge is the lipid challenge, the second meal challenge is the glucose challenge and third meal challenge is the mixed-meal challenge.
  Interventions: Dietary Supplement: Lipid Challenge; Dietary Supplement: Glucose Challenge; Dietary Supplement: Mixed Meal Challenge

INTERVENTIONS:
Dietary Supplement: Lipid Challenge — For the lipid challenge, participants consume 100 grams of a long chain triglyceride emulsion in the form of liquid drink, which is the commercially available brand called Calogen, from Nutricia, Inc.
  Other Names: Calogen
Dietary Supplement: Glucose Challenge — For the glucose challenge, participants consume 75 grams of glucose in 200 milliliters of water, which is the World Health Organization (WHO) recommended drink for the Oral Glucose Tolerance Test.
Dietary Supplement: Mixed Meal Challenge — For the mixed-meal challenge, participants consume 237 milliliters of the Ensure Enlive nutrition drink , which contains 11 grams of fat, 22 grams of sugar and 20 grams of protein.
  Other Names: Ensure Enlive

SUMMARY:
The purpose of this study is to assess sample collection conditions for various dietary challenges (fat, sugar, and mixed) and determine the optimal fasting and post-meal sample collection time points for future studies on a larger group of individuals. Study participants will attend three study visits where they take part in lipid, glucose, and mixed meal challenges. At each of the three visits, participants will provide venous blood samples and a urine sample before consuming the test meal and will provide 6 additional venous finger blood samples post-meal.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading killer of Americans, accounting for more than 800,000 deaths each year. A vital step in reducing the number of heart disease-related deaths in the U.S. is to identify those at probable risk. The Clinical Chemistry Branch (CCB) in the Division of Laboratory Sciences (DLS) at the Centers for Disease Control and Prevention (CDC) has developed advanced analytical methods for assessing the risk for lipid metabolism related diseases, including CVD. This comprehensive analytical method measures levels of protein and lipid constituents of lipoprotein size and density classes (e.g. high-density lipoprotein (HDL), low-density lipoprotein (LDL) and very low-density lipoprotein (VLDL)) in blood. The analytical method uses asymmetric flow-field flow fractionation (AF4) to separate lipoprotein classes (HDL, LDL, VLDL) in serum or plasma into size fractions, and in each fraction quantifies over 50 CVD-linked biomarkers by isotope dilution tandem mass spectrometry. The CCB plans to apply the measurement of this wide array of biomarkers in future epidemiologic investigations of CVD. These studies have the potential to expand the number of diagnostically relevant CVD risk factors that currently are limited to cholesterol and triglyceride measurements.

However, there is limited information about how the CVD-linked biomarkers measured with the CCB's method are affected by blood collection conditions and the fasting/non-fasting state of individuals. Furthermore, lipid metabolism is very dynamic and the absolute levels of biomarkers are strongly affected by each individual's diet, lifestyle, gender, age, and physiology. Thus, assessing biomarkers related to lipid metabolism is most effective in a pre- and post-test comparison (i.e. fasting vs. after a test meal) with controlled lipid and carbohydrate content.

The study involves three different meal challenges on three separate days with approximately two weeks in between. The first meal challenge will involve the consumption of a standardized mixture of dietary fats (lipid challenge), the second meal challenge will be a sugar sweetened beverage (glucose challenge) and the third meal challenge will be a nutrition shake (mixed meal challenge). At each of the three visits, each individual will provide both venous and finger-prick blood samples and a urine sample before consuming the test meal (in a fasting state) and 6 additional venous and finger-prick blood samples post-meal at described intervals. Each study visit will last approximately 8 hours.

ELIGIBILITY:
Inclusion Criteria:

Any adult (18 -50 years) may participate who agrees to complete the following requirements:

* Be functionally ambulatory
* Have a body mass index (BMI) between >20 kg/m2 to <40 kg/m2
* Be available for an 8-hour visit to the Emory University Hospital Clinical Research Center
* Be able to fast for 10 hours prior to visiting Emory University Hospital Clinical Research Unit for each meal challenge

Exclusion Criteria:

* Vulnerable populations which include children, pregnant women, individuals with mental disabilities, and prisoners will be excluded from the study.
* Individuals with history of GI symptoms or fat intolerance will be excluded from the study.
* Individuals with health condition that would put them in risk due to 10 hour fasting, including:

  1. Has taken any diabetic or lipid lowering prescription medications within the past 12 months
  2. History of chronic diseases
  3. Hospitalized within the last year
  4. Currently pregnant
  5. Current active malignant neoplasm or history of malignancy (other than localized basal cell cancer of the skin) during the previous 5 years
  6. Current chronic autoimmune or pro-inflammatory disease
  7. History of tuberculosis, HIV, or other chronic infection
  8. Previous diagnosis of type 1 or type 2 diabetes with active treatment with insulin or other glucose lowering medication
  9. Advanced (>= stage 3) renal disease
  10. Recreational or prescription drug or alcohol abuse
  11. Any history of gastrointestinal diseases, including malabsorption
  12. Any history of intolerance to dietary fat
  13. Inability to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Change in high-density lipoprotein (HDL) Size | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  HDL concentration size profiles for each time-point will be determined for each of the three meal challenges. HDL is considered to be anti- atherogenic because of its ability deplete excess cholesterol accumulating necrotic cores and repair arterial lesions.
Change in low-density lipoprotein (LDL) Size | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  LDL concentration size profiles for each time-point will be determined for each of the three meal challenges. LDL is considered to be atherogenic because it is likely to be trapped inside the intima of blood vessels and arteries and initiate inflammatory response, foam-cell formation, and smooth muscle cell proliferation, leading to development necrotic cores, lesions, plaques and their eventual rupture. Elevated LDL has been thought to contribute to atherosclerotic events, however, research has also observed coronary events occurring in individuals with LDL levels in the acceptable range.
Change in Total Cholesterol | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Total cholesterol profiles for each time-point will be determined for each of the three meal challenges. Elevated total cholesterol has been thought to contribute to atherosclerotic events, however, research has also observed coronary events occurring in individuals with total cholesterol levels in the acceptable range.
Change in Free Cholesterol | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Free cholesterol concentration for each time-point will be determined for each of the three meal challenges. Free cholesterol is unesterified cholesterol that is circulating in the blood stream.
Change in Cholesterol Ester | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Cholesterol ester concentration for each time-point will be determined for each of the three meal challenges. Lipoproteins contain cholesterol ester, and cholesterol ester is associated with atherosclerosis.
Change in Triglycerides | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Triglyceride concentration for each time-point will be determined for each of the three meal challenges. Triglycerides peak in serum 2 to 4 hours after a meal and return to a pre-meal state in 6 to 8 hours.
Change in Phosphatidylinositol | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Phosphatidylinositol concentration for each time-point will be determined for each of the three meal challenges.
Change in Phosphatidylethanolamine | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Phosphatidylethanolamine concentration for each time-point will be determined for each of the three meal challenges.
Change in Phosphatidylcholine | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Phosphatidylcholine concentration for each time-point will be determined for each of the three meal challenges.
Change in Sphingomyelin | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Sphingomyelin concentration for each time-point will be determined for each of the three meal challenges.
Change in Lysophosphatidylcholine | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Lysophosphatidylcholine concentration for each time-point will be determined for each of the three meal challenges.
Change in Apolipoprotein AI | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Apolipoprotein AI concentration for each time-point will be determined for each of the three meal challenges.
Change in Apolipoprotein AII | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Apolipoprotein AII concentration for each time-point will be determined for each of the three meal challenges.
Change in Apolipoprotein AIV | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Apolipoprotein AIV concentration for each time-point will be determined for each of the three meal challenges.
Change in Apolipoprotein B | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Apolipoprotein B concentration for each time-point will be determined for each of the three meal challenges.
Change in Apolipoprotein CI | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Apolipoprotein CI concentration for each time-point will be determined for each of the three meal challenges.
Change in Apolipoprotein CII | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Apolipoprotein CII concentration for each time-point will be determined for each of the three meal challenges.
Change in Apolipoprotein CIII | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Apolipoprotein CIII concentration for each time-point will be determined for each of the three meal challenges.
Change in Apolipoprotein E | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Apolipoprotein E concentration for each time-point will be determined for each of the three meal challenges.
Change in Lecithin-Cholesterol Acyltransferase | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Lecithin-cholesterol acyltransferase concentration for each time-point will be determined for each of the three meal challenges.
Change in Cholesterol Ester Transfer Protein | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Cholesterol ester transfer protein concentration for each time-point will be determined for each of the three meal challenges.
Change in Lipoprotein (a) | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Lipoprotein (a) concentration for each time-point will be determined for each of the three meal challenges.
Change in Phospholipid Transfer Protein | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Phospholipid transfer protein concentration for each time-point will be determined for each of the three meal challenges.
Change in Serum Paraoxonase/arylesterase 1 | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Serum paraoxonase/arylesterase 1 concentration for each time-point will be determined for each of the three meal challenges.
Change in Serum Amyloid A1 | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Serum amyloid A1 concentration for each time-point will be determined for each of the three meal challenges.
Change in Serum Amyloid A4 | Baseline, Minute 15, Minute 30, Hour 1, Hour 2, Hour 4 and Hour 6 during study visits 1, 2, and 3 (up to 6 weeks)
  Serum amyloid A4 concentration for each time-point will be determined for each of the three meal challenges.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ziegler, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT05087823/ICF_000.pdf